CLINICAL TRIAL: NCT01235767
Title: Effect of Animal Source Food Supplement Prior to and During Pregnancy on Birth Weight and Prematurity in Rural Vietnam
Brief Title: Animal Source Food Supplement and Pregnancy in Vietnam
Acronym: VACVINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-068; TRF-01 (Other Grant/Funding Number: Thrasher Research Fund)
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Low Birth Weight; Preterm Birth
Keywords: birth weight; prematurity; gestational age; low birth weight; pregnancy; nutrition; Vietnam
MeSH Terms: conditions — Premature Birth; Birth Weight | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASF supplement pre-pregnancy to term (Experimental): Supplement of animal-source foods rich in iron, zinc, vitamin A, and vitamin B12
  Interventions: Other: Food
- ASF Supplement mid-gestation to term (Experimental): Supplement of animal-source foods rich in iron, zinc, vitamin A, and vitamin B12
  Interventions: Other: Food
- Routine prenatal care (No Intervention): Nutrition education and iron-folate supplements during pregnancy

INTERVENTIONS:
Other: Food — Animal-source food (ASF) supplement rich in iron, zinc, vitamin A, and vitamin B12 taken week-days at mid-morning separate from other food. Length of intervention is either from pre-pregnancy (time of registration to marry) to term or from 16 weeks gestation to term.
  Arms: ASF Supplement mid-gestation to term; ASF supplement pre-pregnancy to term

SUMMARY:
The purpose of this study is to determine if a nutrient-rich supplement of animal-source foods ingested 5d/wk from pre-conception to term improves maternal nutrient status, decreases infections, and improves birth weight and rates of prematurity compared with supplemental ingestion during pregnancy ( from mid-gestation to term) or routine prenatal care.

DETAILED DESCRIPTION:
It has been known for over 80 years that maternal starvation reduces fetal growth and increases neonatal infections. Many different nutrition programs have been targeted to pregnant women to improve pregnancy outcomes. The impact of these programs has been disappointing, and the prevalence of low birth weight (LBW) and infant mortality remains high, especially in developing countries. More recently, as a result of improved access to cereals following the 'green revolution,' nutritional concerns shifted from protein and energy to micronutrient deficiencies, especially those micronutrients in animal-source foods (ASFs)-iron, zinc, vitamins A and B12. Diets of pregnant women are usually limited to rice and a few vegetables, and they lack key nutrients known to reduce preterm delivery, to support fetal growth, and to prevent infections that leads to early neonatal deaths. Vietnam has a well-established farm system that supports the local production of fish, pork, poultry, and eggs. This provides an opportunity to evaluate the impact of a food-based, micronutrient-rich supplement on pregnancy outcome in high-risk, rural Vietnamese women. Since maternal nutritional status at conception is strongly linked to pregnancy outcomes, we will compare the effect of consuming a micronutrient-rich, animal-source food (ASF) supplement from pre-conception to term with a supplement from mid-gestation to term or routine prenatal care on infant birth weight, prematurity rate, and infant growth during the first 6 months of life. This study will be the first to compare a food-based, micronutrient-rich supplement consumed prior to conception to term with one given only during pregnancy. Although it is recognized by many that pregnancy may be too narrow a window to improve maternal nutritional health, it is typical for micronutrient supplements to only be given from the time of enrolling for prenatal care to term. The results of our study, therefore, will have world-wide implications regarding when maternal supplementation should be given to have the greatest impact on pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women registering to marry in the Cam Khe District of Phu Tho Province
* Nulliparous
* Planning to reside in the study site for the next 3 years.

Exclusion Criteria:

* Married
* Have had a previous pregnancy
* Have a history of severe infections (HIV, TB) or metabolic disease (diabetes)
* BMI <17 kg/m2
* Do not reside in study communes
* Unable to provide informed consent

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 291 (Actual)
Dates: Start 2011-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Birth Weight | At birth
  Weight of baby at birth on a scale weighing to 0.1 g made within one hour of delivery

SECONDARY OUTCOMES:
Preterm birth | At birth
  Birth of baby prior to 37 weeks gestation based on mother's last menstrual period, confirmed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Janet C King, Ph.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- National Institute of Nutrition, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quyen PN, Nga HT, Chaffee B, Ngu T, King JC. Effect of maternal prenatal food supplementation, gestational weight gain, and breast-feeding on infant growth during the first 24 months of life in rural Vietnam. PLoS One. 2020 Jun 25;15(6):e0233671. doi: 10.1371/journal.pone.0233671. eCollection 2020. PMID 32584881
- [Derived] Nga HT, Quyen PN, Chaffee BW, Diep Anh NT, Ngu T, King JC. Effect of a nutrient-rich, food-based supplement given to rural Vietnamese mothers prior to and/or during pregnancy on birth outcomes: A randomized controlled trial. PLoS One. 2020 May 29;15(5):e0232197. doi: 10.1371/journal.pone.0232197. eCollection 2020. PMID 32469870